CLINICAL TRIAL: NCT03713632
Title: A Randomized, Double-blind, Multicenter Study Assessing Short (16 Weeks) and Long-term Efficacy (up to 1 Year), Safety, and Tolerability of 2 Subcutaneous Secukinumab Dose Regimens in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (SUNRISE)
Brief Title: Study of Efficacy and Safety of Two Secukinumab Dose Regimens in Subjects With Moderate to Severe Hidradenitis Suppurativa (HS)
Acronym: SUNRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457M2302; 2018-002062-39 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: acne inversa; Hidradenitis suppurativa; maladie de Verneuil; inflammatory disease; AIN457; AIN457M; secukinumab; HS; lumps; skin; lesions
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Secukinumab 1 (Active Comparator): Secukinumab 300mg every 2 weeks
  Interventions: Drug: Secukinumab
- Secukinumab 2 (Active Comparator): Secukinumab 300mg every 4 weeks
  Interventions: Drug: Secukinumab
- Placebo 1 (Placebo Comparator): Placebo group to secukinumab 300mg every 2 weeks
  Interventions: Drug: Placebo
- Placebo 2 (Placebo Comparator): Placebo group to secukinumab 300mg every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300mg every 2 or every 4 weeks
  Arms: Secukinumab 1; Secukinumab 2
Drug: Placebo — Placebo 300mg every 2 or every 4 weeks
  Arms: Placebo 1; Placebo 2

SUMMARY:
The purpose of this study was to demonstrate superiority of secukinumab at Week 16, based on Hidradenitis Suppurativa Clinical Response (HiSCR) rates versus placebo, along with the maintenance of efficacy of secukinumab at Week 52 in subjects with moderate to severe HS. Moreover, this study assessed the safety and tolerability of secukinumab.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled, parallel group study with two secukinumab dose regimens in patients with moderate to severe HS. The study consisted of: screening (up to 4 weeks) treatment period 1 (16 weeks, active drug or placebo) and treatment period 2 (up to 1 year all patients on active drug); there was an optional extension study (NCT04179175). Adult males and females with moderate to severe HS were included, with a diagnosis of HS greater than 1 year prior to baseline. Dosing was once every 2 weeks, or once every 4 weeks via pre-filled syringe; periodic home-dosing is included.

In Treatment Period 1, participants were randomized to secukinumab Q2W, secukinumab Q4W, placebo Q2W or placebo Q4W in 1:1:0.5:0.5 ratio. In Treatment Period 2, at the Week 16 visit participants initially randomized to placebo were switched to one of the two active dose regimens (secukinumab Q2W or Q4W), while subjects randomized to secukinumab during Treatment Period 1 continued on the same dose.

ELIGIBILITY:
Inclusion Criteria:

* -Written informed consent must be obtained before any assessment is performed.
* Male and female patients ≥ 18 years of age.
* Diagnosis of HS ≥ 1 year prior to baseline.
* Patients with moderate to severe HS defined as:
* A total of at least 5 inflammatory lesions, i.e. abscesses and/or inflammatory nodules AND
* Inflammatory lesions should affect at least 2 distinct anatomic areas
* Patients agree to daily use of topical over-the-counter antiseptics on the areas affected by HS lesions while on study treatment.

Exclusion Criteria:

* Total fistulae count ≥ 20 at baseline.
* Any other active skin disease or condition that may interfere with assessment of HS.
* Active ongoing inflammatory diseases other than HS that require treatment with prohibited medications.
* Use or planned use of prohibited treatment. Washout periods detailed in the protocol have to be adhered to.
* History of hypersensitivity to any of the study drug constituents.
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Lead Study Director, Study Director — Novartis
Locations (101):
- United States (14):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Whittier, California
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Sandy Springs, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Bellaire, Texas
  - Novartis Investigative Site, Pflugerville, Texas
  - Novartis Investigative Site, Norfolk, Virginia
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Capital Federal
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Canada (4):
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Richmond Hill, Ontario
  - Novartis Investigative Site, Drummondville, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
- Colombia (2):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Zagreb, HRV, Croatia
- Czechia (2):
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Jihlava
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen NV
- France (9):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Saint-Mandé
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Würzburg
- Greece (2):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (3):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
- India (2):
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Navi Mumbai, Maharashtra
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Saida, Lebanon
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius, Vilniaus
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Johor Bahru
- Novartis Investigative Site, Bergen op Zoom, Netherlands
- Novartis Investigative Site, Makati City, Philippines
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Prešov
- South Africa (2):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Soweto, Gauteng
- Spain (5):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (5):
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, London
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Alavi A, Reguiai Z, Jemec GBE, Gottlieb AB, Wozniak MB, Uhlmann L, Fan H, Llobet Martinez A, Bruin G, Thomas N, Alarcon I, Bieth B, Ravichandran S, Kimball AB. Secukinumab in the Treatment of Moderate-to-Severe Hidradenitis Suppurativa: Pooled Pharmacokinetics and Safety Results From the SUNSHINE and SUNRISE Phase 3 Studies. Int J Dermatol. 2026 Feb;65(2):289-298. doi: 10.1111/ijd.70025. Epub 2025 Aug 21. PMID 40839197
- [Derived] Ingram JR, Szepietowski JC, Matusiak L, Kokolakis G, Wozniak MB, Ortmann CE, Martinez AL, Ravichandran S, Thomas N, Alarcon I, Pieterse CC, Alam MS, Ioannides D, Kimball AB. Assessing Long-Term Pain Reduction with Secukinumab in Moderate to Severe Hidradenitis Suppurativa: A Post Hoc Analysis of the SUNSHINE and SUNRISE Phase 3 Trials. Dermatol Ther (Heidelb). 2025 Jul;15(7):1833-1849. doi: 10.1007/s13555-025-01426-x. Epub 2025 May 15. PMID 40372667
- [Derived] Zouboulis CC, Kyrgidis A, Alavi A, Jemec GBE, Martorell A, Marzano AV, van der Zee HH, Wozniak MB, Martinez AL, Kasparek T, Bachhuber T, Ortmann CE, Lobach I, Thomas N, Ravichandran S, Tzellos T. Secukinumab efficacy in patients with hidradenitis suppurativa assessed by the International Hidradenitis Suppurativa Severity Score System (IHS4): A post hoc analysis of the SUNSHINE and SUNRISE trials. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1421-1430. doi: 10.1111/jdv.20369. Epub 2024 Oct 19. PMID 39425517
- [Derived] Passera A, Muscianisi E, Demanse D, Okoye GA, Jemec GBE, Mayo T, Hsiao J, Shi VY, Byrd AS, Wei X, Uhlmann L, Vandemeulebroecke M, Ravichandran S, Porter ML. New insights on hidradenitis suppurativa phenotypes and treatment response: An exploratory automated analysis of the SUNSHINE and SUNRISE trials. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1410-1420. doi: 10.1111/jdv.20234. Epub 2024 Aug 5. PMID 39101698
- [Derived] Kimball AB, Jemec GBE, Alavi A, Reguiai Z, Gottlieb AB, Bechara FG, Paul C, Giamarellos Bourboulis EJ, Villani AP, Schwinn A, Rueff F, Pillay Ramaya L, Reich A, Lobo I, Sinclair R, Passeron T, Martorell A, Mendes-Bastos P, Kokolakis G, Becherel PA, Wozniak MB, Martinez AL, Wei X, Uhlmann L, Passera A, Keefe D, Martin R, Field C, Chen L, Vandemeulebroecke M, Ravichandran S, Muscianisi E. Secukinumab in moderate-to-severe hidradenitis suppurativa (SUNSHINE and SUNRISE): week 16 and week 52 results of two identical, multicentre, randomised, placebo-controlled, double-blind phase 3 trials. Lancet. 2023 Mar 4;401(10378):747-761. doi: 10.1016/S0140-6736(23)00022-3. Epub 2023 Feb 3. PMID 36746171
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1840

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled in 132 study sites worldwide.
Groups:
- AIN457 Q2W: Secukinumab 300mg every 2 weeks (Treatment Period 1 and 2)
- AIN457 Q4W: Secukinumab 300mg every 4 weeks (Treatment Period 1 and 2)
- Placebo: Placebo group to secukinumab 300mg (Treatment Period 1)
- Placebo - Re-randomized to AIN457 Q2W: Placebo group, re-randomized to secukinumab 300mg Q2W at week 16 (Treatment Period 2)
- Placebo - Re-randomized to AIN457 Q4W: Placebo group, re-randomized to secukinumab 300mg Q4W at week 16 (Treatment Period 2)
Period: Treatment Period 1 (Until Week 16)
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo | Placebo - Re-randomized to AIN457 Q2W | Placebo - Re-randomized to AIN457 Q4W
Started | 181 (1 patient was mis randomized and excluded from the full analysis set.) | 180 | 183 | 0 | 0
Full Analysis Set | 180 | 180 | 183 | 0 | 0
Completed | 170 | 169 | 167 | 0 | 0
Not Completed | 11 | 11 | 16 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 8 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0 | 0
Not completed — Technical problems | 1 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Misrandomized Subject | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (After Week 16)
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo | Placebo - Re-randomized to AIN457 Q2W | Placebo - Re-randomized to AIN457 Q4W
Started | 170 | 169 | 0 | 81 | 86
Completed | 149 | 133 | 0 | 68 | 69
Not Completed | 21 | 36 | 0 | 13 | 17
Not completed — Withdrawal by Subject | 9 | 18 | 0 | 9 | 12
Not completed — Adverse Event | 6 | 3 | 0 | 2 | 1
Not completed — Lack of Efficacy | 3 | 3 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 8 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 2
Not completed — Technical Problems | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- AIN457 Q2W: Secukinumab 300mg every 2 weeks
- AIN457 Q4W: Secukinumab 300mg every 4 weeks
- Placebo: Placebo group to secukinumab 300mg
- Total: Total of all reporting groups
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo | Total
Number analyzed (Participants) | 180 | 180 | 183 | 543
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (11.48) | 35.5 (11.41) | 36.2 (11.25) | 36.3 (11.38)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 177 | 178 | 181 | 536
  >=65 years | 3 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 103 | 105 | 306
  Male | 82 | 77 | 78 | 237
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 133 | 139 | 143 | 415
  Black or African American | 18 | 19 | 12 | 49
  Asian | 16 | 16 | 19 | 51
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  American Indian or Alaska native | 7 | 5 | 8 | 20
  Multiple | 4 | 1 | 1 | 6
  Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hidradenitis Suppurativa Clinical Response (HiSCR50)
Description: HiSCR50 at Week 16 is defined as at least a 50% decrease in Abscess and inflammatory Nodule (AN) count compared to baseline with no increase in the number of abscesses and/or in the number of draining fistulas from baseline to Week 16. The baseline is defined as the last assessment (including unscheduled visits) obtained before/on the day of the first administration of the study treatment, or on the randomization date if there had been no drug administration.
  This endpoint was analyzed by logistic regression.
Time Frame: 16 weeks
Population: Full analysis set (FAS): consisted of all subjects to whom study treatment had been assigned, excluding mis-randomized patients.
  Subjects were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo
Number analyzed (Participants) | 180 | 180 | 183
Percentage of Participants | 42.3 | 46.1 | 31.2
Statistical Analysis 1: Comparison: AIN457 Q2W vs Placebo; Test type: Superiority; p = 0.0149, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.05 to 2.55]
Statistical Analysis 2: Comparison: AIN457 Q4W vs Placebo; Test type: Superiority; p = 0.0022, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.22 to 2.96]

2. Secondary Outcome: Percentage Change From Baseline in AN Count
Description: Percent change from baseline in abscesses and inflammatory nodules (AN) count. This endpoint was analyzed by analysis of covariance.
Time Frame: Baseline, 16 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo
Number analyzed (Participants) | 180 | 180 | 183
Percentage change from baseline | -39.3 (4.43) | -45.5 (4.08) | -22.4 (4.84)
Statistical Analysis 1: Comparison: AIN457 Q2W vs Placebo; Test type: Superiority; p = 0.0051, ANCOVA — one-side p-value; Mean Difference (Net) = -16.33, 95% CI 2-sided [-28.79 to -3.88]
Statistical Analysis 2: Comparison: AIN457 Q4W vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA — one-side p-value; Mean Difference (Net) = -22.94, 95% CI 2-sided [-35.24 to -10.63]

3. Secondary Outcome: Percentage of Participants With Hidradenitis Suppurativa (HS) Flares
Description: Percentage of participants who experience at least one flare over 16 weeks. A flare is defined as at least a 25% increase in abscesses and inflammatory nodules (AN) count with a minimum increase of 2 AN relative to baseline.
  This endpoint was analyzed by logistic regression.
Time Frame: 16 weeks
Population: Full Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo
Number analyzed (Participants) | 180 | 180 | 183
Percentage of Participants | 20.1 | 15.6 | 27.0
Statistical Analysis 1: Comparison: AIN457 Q2W vs Placebo; Test type: Superiority; p = 0.0732, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.41 to 1.14]
Statistical Analysis 2: Comparison: AIN457 Q4W vs Placebo; Test type: Superiority; p = 0.0049, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.29 to 0.84]

4. Secondary Outcome: Percentage of Participants Achieving NRS30
Description: Patients achieving Numerical Rating Scale score of 30 (NRS30) at week 16, defined as at least a 30% reduction and at least one unit reduction from baseline in the Patient's Global assessment of Skin Pain (where range 0 [no skin pain] to 10 [worst skin pain]).
  This endpoint was analyzed by logistic regression.
Time Frame: 16 weeks
Population: Full Analysis Set restricted to participants with baseline NRS score greater or equal to 3
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo
Number analyzed (Participants) | 135 | 129 | 132
Percentage of participants | 38.6 | 34.7 | 22.4
Statistical Analysis 1: Comparison: AIN457 Q2W vs Placebo; Test type: Superiority; p = 0.0026, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.28 to 4.09]
Statistical Analysis 2: Comparison: AIN457 Q4W vs Placebo; Test type: Superiority; p = 0.0206, Regression, Logistic — one-sided p-value; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.03 to 3.37]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from first dose of study treatment, up to approximately 52 weeks for AIN457 (up to 60 weeks for subjects who did not move to the extension study) and up to 16 weeks for placebo.
Description: AEs are any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Groups:
- AIN457 Q2W: Subjects who were randomized to AIN457 (secukinumab) 300mg Q2W dose regimen at the study entry. Adverse events were assessed up to Week 60
- AIN457 Q4W: Subjects who were randomized to AIN457 (secukinumab) 300mg Q4W dose regimen at the study entry. Adverse events were assessed up to Week 60
- Placebo: Subjects who were randomized to matching placebo at the study entry. Adverse events were assessed up to Week 16
- Any AIN457 Q2W: Subjects who received at least 1 dose of secukinumab 300 mg Q2W dose (including subjects who switched from placebo to secukinumab Q2W at Week 16). Adverse events were assessed up to Week 60
- Any AIN457 Q4W: Subjects who received at least 1 dose of secukinumab 300 mg Q4W dose (including subjects who switched from placebo to secukinumab Q4W at Week 16). Adverse events were assessed up to Week 60
- Any AIN457: Subjects who received at least 1 dose of secukinumab
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo | Any AIN457 Q2W | Any AIN457 Q4W | Any AIN457
All-Cause Mortality (participants affected / at risk) | 0/180 | 1/180 | 0/183 | 0/261 | 2/266 | 2/527
Serious Adverse Events (participants affected / at risk) | 19/180 | 15/180 | 5/183 | 22/261 | 23/266 | 45/527
Other Adverse Events (participants affected / at risk) | 123/180 | 125/180 | 84/183 | 174/261 | 174/266 | 348/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2W (N=180) | AIN457 Q4W (N=180) | Placebo (N=183) | Any AIN457 Q2W (N=261) | Any AIN457 Q4W (N=266) | Any AIN457 (N=527)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 1 | 2 | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Unevaluable event (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Amyloidosis (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Colonic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Scrotal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sweat gland infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 0 | 2
Glomerular vascular disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 2
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Scrotal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 5 | 0 | 5
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2W (N=180) | AIN457 Q4W (N=180) | Placebo (N=183) | Any AIN457 Q2W (N=261) | Any AIN457 Q4W (N=266) | Any AIN457 (N=527)
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 2 | 5 | 10 | 15
Abdominal pain upper (Gastrointestinal disorders) | 3 | 9 | 1 | 4 | 10 | 14
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 4 | 1 | 5
Dental caries (Gastrointestinal disorders) | 4 | 1 | 0 | 4 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 13 | 14 | 13 | 19 | 19 | 38
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4 | 1 | 7 | 6 | 13
Haemorrhoids (Gastrointestinal disorders) | 1 | 5 | 0 | 1 | 5 | 6
Nausea (Gastrointestinal disorders) | 6 | 5 | 4 | 12 | 7 | 19
Toothache (Gastrointestinal disorders) | 6 | 5 | 0 | 7 | 5 | 12
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 6 | 1 | 7
Fatigue (General disorders) | 4 | 6 | 2 | 7 | 7 | 14
Influenza like illness (General disorders) | 1 | 5 | 0 | 1 | 5 | 6
Pyrexia (General disorders) | 7 | 8 | 3 | 9 | 12 | 21
Bronchitis (Infections and infestations) | 5 | 5 | 2 | 5 | 7 | 12
COVID-19 (Infections and infestations) | 10 | 7 | 3 | 13 | 14 | 27
Conjunctivitis (Infections and infestations) | 4 | 6 | 0 | 4 | 7 | 11
Ear infection (Infections and infestations) | 4 | 1 | 0 | 5 | 1 | 6
Folliculitis (Infections and infestations) | 9 | 2 | 3 | 9 | 4 | 13
Influenza (Infections and infestations) | 5 | 1 | 0 | 7 | 1 | 8
Nasopharyngitis (Infections and infestations) | 21 | 18 | 16 | 28 | 25 | 53
Oral candidiasis (Infections and infestations) | 5 | 1 | 0 | 5 | 3 | 8
Pharyngitis (Infections and infestations) | 3 | 6 | 3 | 4 | 9 | 13
Rhinitis (Infections and infestations) | 4 | 4 | 1 | 6 | 7 | 13
Sinusitis (Infections and infestations) | 3 | 3 | 3 | 7 | 3 | 10
Skin candida (Infections and infestations) | 6 | 4 | 1 | 8 | 4 | 12
Sweat gland infection (Infections and infestations) | 3 | 2 | 3 | 9 | 2 | 11
Tonsillitis (Infections and infestations) | 2 | 4 | 0 | 4 | 5 | 9
Upper respiratory tract infection (Infections and infestations) | 13 | 8 | 7 | 16 | 11 | 27
Urinary tract infection (Infections and infestations) | 7 | 7 | 5 | 8 | 12 | 20
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 1 | 5 | 6
Gamma-glutamyltransferase increased (Investigations) | 5 | 1 | 0 | 5 | 1 | 6
Lipase increased (Investigations) | 3 | 7 | 1 | 5 | 7 | 12
SARS-CoV-2 test positive (Investigations) | 3 | 4 | 3 | 5 | 4 | 9
Weight decreased (Investigations) | 0 | 4 | 0 | 0 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 5 | 11 | 9 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 12 | 4 | 7 | 14 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3 | 4 | 6 | 10
Dizziness (Nervous system disorders) | 4 | 7 | 3 | 6 | 7 | 13
Headache (Nervous system disorders) | 31 | 27 | 16 | 39 | 36 | 75
Depression (Psychiatric disorders) | 6 | 5 | 4 | 6 | 5 | 11
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 5 | 0 | 3 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 3 | 6 | 9 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 1 | 8 | 9 | 17
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 4 | 4 | 8
Eczema (Skin and subcutaneous tissue disorders) | 10 | 6 | 1 | 11 | 7 | 18
Hidradenitis (Skin and subcutaneous tissue disorders) | 21 | 23 | 14 | 26 | 31 | 57
Intertrigo (Skin and subcutaneous tissue disorders) | 4 | 5 | 0 | 6 | 8 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 3 | 5 | 11 | 5 | 16
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 4 | 0 | 6 | 6 | 12
Hypertension (Vascular disorders) | 11 | 6 | 2 | 14 | 7 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03713632/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03713632/SAP_002.pdf